CLINICAL TRIAL: NCT06717542
Title: Tissue Analysis (Histological, Ultrastructural and Molecular) of Liver Grafts as a Predictor of Transplant Outcome.
Brief Title: Tissue Analysis of Liver Grafts as a Predictor of Transplant Outcome.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: donorHOPE_2022; RC-2022-2773274 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2024-12-01; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Hepatic Transplantation; Rejection; Transplant, Liver
Keywords: Transplant; Liver
MeSH Terms: conditions — Rejection, Psychology | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Intervention Model Description: Two arm designed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Organ donors (Other): organ donors (legally deceased, brain death or cardiac death)
  Interventions: Diagnostic Test: histochemical and immunohistochemical analysis; Diagnostic Test: RT-PCR
- Organ recipients (Other): Organ recipients
  Interventions: Diagnostic Test: histochemical and immunohistochemical analysis; Diagnostic Test: RT-PCR

INTERVENTIONS:
Diagnostic Test: histochemical and immunohistochemical analysis — 2 µm sections will be cut from the paraffin blocks for histochemical and immunohistochemical (IHC) investigations. IHC will be performed with an automated stainer (Ventana/Roche®, Ventana Medical Systems, USA) for the endothelial markers CD34, ERG, Nestin and Caveolin-1
Diagnostic Test: RT-PCR — Custom RT-PCR analyses will be performed manually for the transcripts (mRNA) of the ERG, Nestin, VEGFR and other genes, at the Pathology Anatomy lab hall. 18 (Prof. D'Errico). Total RNA will be extracted from the paraffin blocks with the RecoverAll™ Total Nucleic Acid Isolation kit (Invitrogen). Reverse Transcriptase will be performed with the High Capacity Reverse Transcription kit (Life Technologies), using the specific primers. Real-Time PCR will be performed with the CFX Connect Real-Time PCR Identification System (BioRad).

SUMMARY:
Despite the good clinical results in terms of outcome with the application of HOPE prior to liver transplantation, very little is still known about the phenotypic and molecular changes that occur during perfusion/preservation during HOPE, particularly with regard to endothelial trophism and activation. Delving into these aspects would be very useful to allow personalised perfusion treatments in the future, thus improving the outcome of transplantation.

DETAILED DESCRIPTION:
The primary aim of the study is the identification of specific 'endothelial signatures' (markers on tissue with immunohistochemistry and gene expression with RT-PCR) in liver grafts after HOPE treatment, predictive of transplant outcome. Interventional study without drug, including two cohorts of patients: (1) liver donors, on whom an allocation biopsy for organ quality will be performed (as standard of care); (2) liver recipients (from donors in cohort 1) on whom a study-specific biopsy will be performed as soon as the transplant has taken place (after vascular anastomoses with organ revascularisation). The study-specific biopsy constitutes the intervention of the study; patients will be treated according to the judgement of the physician and the information reported in the Technical Data Sheet of each product of any concomitant therapies administered according to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* For Donors:

Availability of enough tissue for histological, immunohistochemical and RT-PCR analysis.

* HOPE performed on the liver graft prior to transplantation.
* For Recipients:
* Availability of enough tissue for histological, immunohistochemical and RT-PCR analysis.
* Age greater than/equal to 18 years.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Identification of specific '"endothelial signatures" | Within 24 months
  Main outcomes to assess the outcome of transplantation will be the percentage of early (PNF and EAD, within 1 week after transplantation) and late (rejection and complications) complications, as well as mortality among recipients within 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Vasuri, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No